CLINICAL TRIAL: NCT03393052
Title: Left Radial comparEd to Femoral Approach for CORonary Angiography in Patients With Previous CABG StuDy
Acronym: L-RECORD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Collaborators: Korgialenio-Benakio Red Cross Hospital (Other); University General Hospital of Heraklion (Other); AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Tsigkas Grigorios, Interventional Cardiologist, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5602
Record Dates: First submitted 2017-12-31; First posted 2018-01-08 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease; Vascular Access Complication
Keywords: L-RECORD; Radial; Femoral; CABG; coronary artery bypass graft
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Radial access (Active Comparator): Left Radial approach for coronary angiography in patients with prior history of CABG surgery
  Interventions: Procedure: Coronary Angiography
- Femoral access (Active Comparator): Femoral approach for coronary angiography in patients with prior history of CABG surgery
  Interventions: Procedure: Coronary Angiography

INTERVENTIONS:
Procedure: Coronary Angiography — Comparison of left radial versus femoral access during coronary angiography of patients who have undergone coronary artery bypass grafting surgery

SUMMARY:
This randomized, multicenter, prospective study seeks to compare left radial and femoral access during cardiac catheterization of patients with prior history of CABG surgery, with the primary objective of demonstrating that the two access techniques do not differ in the net procedure time (non-inferiority study) expanding the documented benefits of radial access to this group of patients.

DETAILED DESCRIPTION:
Patients from 4 different centers with a history of CABG are randomized 1:1 to left radial or femoral access. Based on the literature, a randomized study sample of a total of 150 patients was calculated with assumptions of 30 +/- 10-minute duration of the procedure, alpha = 5%, beta = 10% (power 90%) and non-inferiority limit Δ = 5 minutes. The primary endpoint of the study is the time it takes after placing the sheath at the initial puncture site until the completion of the diagnostic procedure (Net procedure time). Secondary endpoints include total time of the procedure, fluoroscopy time, total patient exposure radiation, amount of contrast used, possible vascular complications, major cardiovascular events and need for crossover access site.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Written informed consent
3. Clinical indication for coronary angiography in a patient with prior history of CABG
4. Left radial artery has not been used as a graft during CABG

Exclusion Criteria:

1. Age over 90 years
2. Patient's refusal to participate in the study
3. Hemodynamic instability of the patient
4. Failure to place a sheath at the randomization access site
5. Arteriovenous fistula at the left upper limb
6. Use of right internal mammary artery as a graft during CABG
7. Creatinine clearance <30 ml/min

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Net Procedure Time | 24 hours
  The time (min) after placement of the sheath at the initial puncture site until the completion of the diagnostic coronary angiography

SECONDARY OUTCOMES:
Total Procedure Time | 24 hours
  The time (min) from local anesthesia at the access site until the completion of the diagnostic coronary angiography
Fluoroscopy Time | 24 hours
  Radiation time (min) after placing the sheath at the initial puncture site until the completion of the diagnostic coronary angiography
Dose Area Product | 24 hours
  Radiation DAP (mGy*cm2) during the diagnostic coronary angiography
Contrast Volume | 24 hours
  Contrast volume (ml) used during the diagnostic coronary angiography
Crossover access site | 24 hours
  Need for crossover access site, other than this of randomization
Major Cardiovascular Events | 24 hours
  Death, stroke, acute myocardial infarction
Vascular Complications | 24 hours
  Vascular access complications

CONTACTS AND LOCATIONS:
Overall Officials: George Hahalis, Prof., Study Director — University Hospital of Patras; Periklis Davlouros, Ass. Prof., Study Director — University Hospital of Patras; Grigorios Tsigkas, Principal Investigator — University Hospital of Patras; Athanasios Makris, Principal Investigator — University Hospital of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pancholy SB, Joshi P, Shah S, Rao SV, Bertrand OF, Patel TM. Effect of Vascular Access Site Choice on Radiation Exposure During Coronary Angiography: The REVERE Trial (Randomized Evaluation of Vascular Entry Site and Radiation Exposure). JACC Cardiovasc Interv. 2015 Aug 17;8(9):1189-1196. doi: 10.1016/j.jcin.2015.03.026. Epub 2015 Jul 22. PMID 26210808
- [Background] Koltowski L, Koltowska-Haggstrom M, Filipiak KJ, Kochman J, Golicki D, Pietrasik A, Huczek Z, Balsam P, Scibisz A, Opolski G. Quality of life in patients with ST-segment elevation myocardial infarction undergoing percutaneous coronary intervention--radial versus femoral access (from the OCEAN RACE Trial). Am J Cardiol. 2014 Aug 15;114(4):516-21. doi: 10.1016/j.amjcard.2014.05.030. Epub 2014 Jun 6. PMID 25015695
- [Background] Michael TT, Alomar M, Papayannis A, Mogabgab O, Patel VG, Rangan BV, Luna M, Hastings JL, Grodin J, Abdullah S, Banerjee S, Brilakis ES. A randomized comparison of the transradial and transfemoral approaches for coronary artery bypass graft angiography and intervention: the RADIAL-CABG Trial (RADIAL Versus Femoral Access for Coronary Artery Bypass Graft Angiography and Intervention). JACC Cardiovasc Interv. 2013 Nov;6(11):1138-44. doi: 10.1016/j.jcin.2013.08.004. Epub 2013 Oct 16. PMID 24139930
- [Background] Louvard Y, Lefevre T, Allain A, Morice M. Coronary angiography through the radial or the femoral approach: The CARAFE study. Catheter Cardiovasc Interv. 2001 Feb;52(2):181-7. doi: 10.1002/1522-726x(200102)52:23.0.co;2-g. PMID 11170325
- [Background] Koutouzis M, Matejka G, Olivecrona G, Grip L, Albertsson P. Radial vs. femoral approach for primary percutaneous coronary intervention in octogenarians. Cardiovasc Revasc Med. 2010 Apr-Jun;11(2):79-83. doi: 10.1016/j.carrev.2009.04.107. PMID 20347796
- [Background] Baker NC, O'Connell EW, Htun WW, Sun H, Green SM, Skelding KA, Blankenship JC, Scott TD, Berger PB. Safety of coronary angiography and percutaneous coronary intervention via the radial versus femoral route in patients on uninterrupted oral anticoagulation with warfarin. Am Heart J. 2014 Oct;168(4):537-44. doi: 10.1016/j.ahj.2014.06.016. Epub 2014 Jul 3. PMID 25262264
- [Background] Jolly SS, Yusuf S, Cairns J, Niemela K, Xavier D, Widimsky P, Budaj A, Niemela M, Valentin V, Lewis BS, Avezum A, Steg PG, Rao SV, Gao P, Afzal R, Joyner CD, Chrolavicius S, Mehta SR; RIVAL trial group. Radial versus femoral access for coronary angiography and intervention in patients with acute coronary syndromes (RIVAL): a randomised, parallel group, multicentre trial. Lancet. 2011 Apr 23;377(9775):1409-20. doi: 10.1016/S0140-6736(11)60404-2. Epub 2011 Apr 4. PMID 21470671
- [Background] Jolly SS, Amlani S, Hamon M, Yusuf S, Mehta SR. Radial versus femoral access for coronary angiography or intervention and the impact on major bleeding and ischemic events: a systematic review and meta-analysis of randomized trials. Am Heart J. 2009 Jan;157(1):132-40. doi: 10.1016/j.ahj.2008.08.023. Epub 2008 Nov 1. PMID 19081409